CLINICAL TRIAL: NCT04988464
Title: A Randomized Controlled Trial of Sleep Scholar: A Single-Session, Internet-Based Insomnia Intervention for College Students
Brief Title: A Single-Session Online Insomnia Intervention
Acronym: SSIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Collaborators: Military Suicide Research Consortium (Other)
Responsible Party: Principal Investigator, Eric Crosby, Principal Investigator, Auburn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #20-555
Record Dates: First submitted 2021-07-08; First posted 2021-08-03 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Insomnia
Keywords: insomnia; suicide prevention; intervention; college students
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Suicide Prevention

STUDY DESIGN:
Intervention Model Description: Participants will complete at least five daily sleep diaries over one week, complete a pre-treatment survey assessment, be randomized in a 1:1 manner into either Sleep Scholar or Building Healthy Habits, complete a post-treatment survey assessment, then complete at least five daily sleep diaries each week for four weeks, and complete a survey assessment both one-week and one-month post-treatment. In total, participants will complete daily sleep diaries for five weeks (35 days) and survey assessments pre-treatment, post-treatment, one-week post-treatment, and one-month post-treatment.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Scholar (Experimental): Sleep Scholar is a fully automated, single-session, self-guided, internet-based CBT-I intervention that participants will read from a web browser on their electronic device. Sleep Scholar's content was adapted from Ellis and colleague's, Morin's, and Perlis and colleague's protocols for therapist-guided CBT-I interventions. Sleep Scholar will be completed in approximately 30 minutes and consists of three successive text-based modules: Sleep Education, Initiating Sleep, and Enhancing Sleep Quality. New content (e.g., vignettes and quizzes) was created to tailor the intervention to college students. For example, after each module, short multiple choice and/or true-false question will be administered to assess participants' understanding of Sleep Scholar's strategies. Participants will be automatically provided feedback on their responses to ensure their understanding of Sleep Scholar's strategies.
  Interventions: Behavioral: Sleep Scholar
- Building Healthy Habits (Placebo Comparator): Building Healthy Habits will be used as the control condition. It combines two modules being utilized as the control condition in an ongoing randomized controlled trial. It is a single-session, self-guided, internet-based intervention that participants will read from a web browser on their electronic device. Building Healthy Habits was piloted by undergraduate research assistants to ensure that it was approximately the same duration as Sleep Scholar (i.e., 30 minutes). It consists of two successive text-based modules focused on healthy movement and healthy eating.
  Interventions: Behavioral: Building Healthy Habits

INTERVENTIONS:
Behavioral: Sleep Scholar — A single-session, internet-based insomnia intervention for college students
  Arms: Sleep Scholar
Behavioral: Building Healthy Habits — A single-session, self-guided, internet-based intervention focused on healthy eating and exercise
  Arms: Building Healthy Habits

SUMMARY:
Cognitive-Behavioral Therapy for Insomnia (CBT-I) is a promising suicide intervention for college students because insomnia is robust risk factor for suicide ideation and CBT-I reduces suicide ideation. Moreover, CBT-I can be self-guided and internet-based, brief, and relatively lower in stigma compared to treatment specifically targeting suicide ideation. However, self-guided, internet-based CBT-I is not brief, and brief CBT-I is neither self-guided nor internet-based. In addition, CBT-I is not usually designed to address the unique experiences of college students. Therefore, this study is a randomized-controlled trial examining the efficacy of Sleep Scholar, a single-session, internet-based insomnia intervention tailored to the needs of college students. The investigators hypothesize that Sleep Scholar will improve insomnia, sleep diary variables (e.g., sleep latency), sleep quality, dysfunctional beliefs about sleep, suicide ideation, depressive, anxiety, and PTSD symptoms over time and compared to a control condition (Building Healthy Habits). The investigators will recruit college students with at least subclinical insomnia symptoms. Participants will complete seven daily pre-treatment sleep diaries and a pre-treatment assessment then be randomized to either Sleep Scholar or Building Healthy Habits, the control single-session, internet-based health intervention condition. After the intervention, participants will complete a post-treatment assessment of acceptability and satisfaction, implement the intervention's strategies, and complete daily sleep diaries for the following four weeks. In addition, participants will complete a one-week and one-month follow-up. If found to be efficacious, Sleep Scholar has the potential to be widely disseminated to college students with insomnia symptoms.

DETAILED DESCRIPTION:
In 2019, college-aged adults in the United States (18-25-year-olds) had the highest rate of past-year suicide ideation (11.8%) compared to any other age group. In addition, the rate of suicide ideation among college-aged adults in the United States has been rising in recent years, especially during the COVID-19 pandemic. Despite the need for mental health treatment among college students, only approximately half of college students experiencing suicide ideation received treatment in the past year, reporting limited access to mental health treatment due to time constraints, financial costs, stigma, concerns about privacy, and an inconvenient location of treatment facilities. Insomnia treatment is a particularly promising target for suicide prevention efforts among college students because insomnia is fairly common, insomnia is a robust risk factor for suicide ideation, and insomnia treatments improve suicide ideation. Moreover, insomnia treatments can be self-guided and internet-based, brief, and relatively lower in stigma compared to treatment specifically targeting suicide ideation. However, current self-guided, internet-based insomnia treatments require a time-intensive process, and current brief insomnia treatments require a trained professional. In addition, previous randomized controlled trials that examined the efficacy of insomnia treatment have recruited samples that are mostly older than college-aged adults and the interventions were not developed with the unique sleep needs of college students in mind. As such, the generalizability of insomnia treatments to college students is unknown. Therefore, the current study aims to examine the efficacy of Sleep Scholar, a single-session, internet-based insomnia intervention tailored to the needs of college students with at least subclinical insomnia symptoms and a lifetime history of suicide ideation.

Insomnia

Approximately 10% of college students meet criteria for insomnia disorder, and approximately one-third of college students have subclinical insomnia symptoms. College students experience a variety of stressors, including transitioning to a new environment, interpersonal difficulties (e.g., family and romantic partners), and increased academic responsibilities. These stressful life events may increase their risk for developing insomnia symptoms through poor sleep hygiene. For example, college students commonly report experiencing noise from roommates and neighbors in the hallway when attempting to sleep and an uncomfortable bedroom temperature as they may not be able to control their dorm room's temperature or may have a difference temperature preference from their roommate. In addition, college-aged adults are significantly more likely to use electronic devices (e.g., cell phone, laptop, video games) before attempting to sleep compared to middle-aged and older adults. College-aged adults are also more like to engage in binge drinking and misuse of stimulant medication compared to middle-aged or older adults. Furthermore, compared with middle-aged and older adults, college students report a greater discrepancy between their weekday and weekend sleep patterns, possibly due to staying up late to socialize with friends. This may be why college students with insomnia spend a greater amount of time in bed and have greater variability in their sleep-wake schedule compared to adults with insomnia that are older.

Insomnia and Mental Health Conditions

Insomnia symptoms are a transdiagnostic factor for other common mental health conditions. Among individuals with insomnia disorder, almost one-third (32%) report suicide ideation. Two meta-analyses showed that insomnia had a positive relationship with suicide ideation. This relationship held across cross-sectional and longitudinal designs, various populations, and while controlling for covariates (e.g., depression and anxiety). In addition, two longitudinal studies included in the meta-anylses showed that the relationship between insomnia and suicide ideation is unidirectional, where insomnia predicted subsequent suicide ideation, but the reverse was not true. Last, in both meta-analyses, insomnia had the strongest and most consistent relationship with suicide ideation compared to the other sleep disturbances. Similarly, approximately 7 to 12% of college students experience depressive, anxiety, and post-traumatic stress disorder (PTSD) symptoms. A meta-analysis of longitudinal studies demonstrated that insomnia symptoms were a positive predictor of depressive and anxiety symptoms, and, a longitudinal study showed that insomnia symptoms were a positive predictor of PTSD symptoms.

Insomnia Interventions

Cognitive-behavioral therapy for insomnia (CBT-I) is a non-pharmacological, evidence-based treatment shown to improve quality and quantity of sleep. Beyond insomnia symptoms, CBT-I improves suicide ideation, depression, anxiety, and PTSD symptoms. There have been several adaptations of traditional CBT-I, including self-guided, internet-based CBT-I and brief, face-to-face CBT-I. Regarding brief, face-to-face CBT-I, when determining the optimal dose of CBT-I, results showed only the one- and four-session conditions significantly improved insomnia symptoms compared to a waitlist control condition. In addition, the single session of CBT-I produced greater positive changes in sleep diary total wake time and sleep efficiency (i.e., proportion of the time in bed that one is sleep) compared to four sessions of CBT-I. Despite the promising evidence that self-guided, internet-based and brief, face-to-face CBT-I interventions reduce suicide ideation and other mental health conditions, self-guided, internet-based CBT-I interventions require a time-intensive process, typically taking several weeks to complete treatment. In addition, there are relatively few single-session CBT-I interventions, and existing single-session CBT-I interventions are not self-guided or internet-based, requiring financial resources and a specific time or location to complete the intervention with a trained professional. Moreover, previous randomized controlled trials that examined the efficacy of insomnia treatment have recruited samples that are mostly older than college-aged adults and the interventions were not developed with the unique sleep needs of college students in mind.

Pilot of Sleep Scholar

Sleep Scholar is a single-session, self-guided, internet-based CBT-I intervention targeted specifically for college students. As such, it has the combined accessibility benefits of both self-guided, internet-based and brief CBT-I interventions. It is accessed through a web browser and completed in approximately 30 minutes without the direct aid of a research assistant or therapist. Sleep Scholar includes three text-based modules based of Psychoeducation, Stimulus Control, and Sleep Quality Enhancement. These modules contain strategies to help college students decrease their excessive time in bed and develop a consistent sleep-wake pattern, including a specific time in bed recommendation. In addition, Sleep Scholar provides vignettes of college students in real-life situations addressing environmental factors, electronic devices before bed, and substance use to improve their insomnia symptoms.

Based on the results of Crosby and Witte's pilot study, several modifications were made to Sleep Scholar based on the Persuasive Systems Design Model of internet-based interventions. Changes were made to support implementation of Sleep Scholar's strategies (e.g., reduced psychological jargon; provided daily sleep diaries while implementing treatment strategies and automatically calculated time in bed adjustments), increase adherence (e.g., access to a website with potential barriers and solutions; during the intervention, asked participants to consider how they will implement difficult goals), and reduce attrition (e.g., sent reminders with loss-framed messages if actions aren't completed by a specific deadline). In addition, reminders were scheduled based on the sleep patterns of participants in the pilot study.

Method

Participants

All study procedures have been approved by the Auburn University Institutional Review Board. Undergraduate students will be recruited from Auburn University using the SONA Human Subject Pool Software and public advertisements. Potential participants will complete an eligibility screener with the inclusion criteria of at least subclinical insomnia (i.e., score ≥8 on the Insomnia Severity Index).

Procedures

Eligible participants will complete an informed consent session with a research assistant via a secure Zoom link. After the consent session, participants will receive text message reminders each morning to complete seven daily sleep diaries. Once participants complete at least five daily sleep diaries, they will be administered a pre-treatment assessment and be randomized in a 1:1 manner into either Sleep Scholar, a single-session, self-guided, internet-based insomnia intervention, or Building Healthy Habits, a single-session, self-guided, internet-based control intervention focused on healthy eating and exercise. Immediately after completing each intervention, participants will complete a post-treatment assessment.

The day after completing the intervention, participants will receive an email that summarizes the key strategies of the intervention and begin receiving daily text message reminders each morning to complete daily sleep diaries for four weeks (28 days). At the end of each week of sleep diaries, sleep diary data will automatically be averaged, and all participants will be provided individualized feedback on their sleep diary variables (e.g., average bedtime and sleep efficiency). However, only participants assigned to Sleep Scholar will be presented their time in bed window recommendation for the next week. In addition, one week and one month after the intervention, all participants will complete a follow-up assessment. In total, participants will complete daily sleep diaries for five weeks (35 days) and survey assessments pre-treatment, post-treatment, one-week post-treatment, and one-month post-treatment.

Hypothesis and Data Analytic Strategy

I hypothesize that Sleep Scholar will improve insomnia, sleep diary variables (e.g., sleep latency), sleep quality, dysfunctional beliefs about sleep, suicide ideation, depressive, anxiety, and PTSD symptoms over time and compared to Building Healthy Habits. All analyses will be based on intention-to-treat. Missing data will be handled with multiple imputation, and all analyses will be conducted with IBM SPSS Statistics (Version 26). The primary outcomes of the intervention's effect on the sleep-related symptoms and secondary outcomes of mental health symptoms will be examined using a 2 x 3 mixed-model repeated measures ANOVA; and sleep diary variables will be examined with a 2 x 5 mixed-model repeated measures ANOVA. ANOVA factors will be condition (i.e., Sleep Scholar and Building Healthy Habits), time (i.e., pre-treatment, one-week follow-up, and one-month follow-up; or weekly averages from the five weeks of daily sleep diaries), and the condition-by-time interaction.

ELIGIBILITY:
Inclusion Criteria:

* At least subclinical insomnia
* Auburn University undergraduate students

Exclusion Criteria:

* Under age 18
* Engagement in shift work
* Untreated restless leg syndrome
* Untreated sleep apnea
* Untreated chronic pain
* Current engagement in insomnia treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
Insomnia | Change from baseline Insomnia Severity Index at one week and one month
  Insomnia Severity Index; range: 0-28; higher score is greater insomnia severity
Sleep Latency | Change from average baseline Sleep Latency at one week, two weeks, three weeks, and four weeks
  The Consensus Sleep Diary; seven daily sleep diaries
Number Of Nocturnal Awakenings | Change from average baseline Number Of Nocturnal Awakenings at one week, two weeks, three weeks, and four weeks
  The Consensus Sleep Diary; seven daily sleep diaries
Duration Of Awakenings After Sleep Onset | Change from average baseline Duration Of Awakenings After Sleep Onset at one week, two weeks, three weeks, and four weeks
  The Consensus Sleep Diary; seven daily sleep diaries
Duration Of Early Morning Awakenings | Change from average baseline Duration Of Early Morning Awakenings at one week, two weeks, three weeks, and four weeks
  The Consensus Sleep Diary; seven daily sleep diaries
Sleep Efficiency | Change from average baseline Sleep Efficiency Index at one week, two weeks, three weeks, and four weeks
  The Consensus Sleep Diary; seven daily sleep diaries; total sleep time divided by total time in bed
Sleep Quality | Change from baseline Pittsburgh Sleep Quality Index at one week and one month
  The Pittsburgh Sleep Quality Index; range: 0-30; higher score is poorer sleep quality
Beliefs and Attitudes About Sleep | Change from baseline Dysfunctional Beliefs and Attitudes about Sleep Scale at one week and one month
  The Dysfunctional Beliefs and Attitudes about Sleep Scale; range: 0-10; higher score is greater dysfunctional beliefs and attitudes about sleep

SECONDARY OUTCOMES:
Suicide Ideation | Change from baseline Depression Symptom Inventory-Suicide Subscale at one week and one month
  Depression Symptom Inventory-Suicide Subscale
Depression | Change from baseline Depression Anxiety Stress Scale - Depression subscale at one week and one month
  The Depression Anxiety Stress Scale - Depression subscale
Anxiety | Change from baseline Depression Anxiety Stress Scale - Anxiety subscale at one week and one month
  The Depression Anxiety Stress Scale - Anxiety subscale
Posttraumatic Stress | Change from baseline Posttraumatic Stress Disorder Checklist for DSM-5 at one week and one month
  The Posttraumatic Stress Disorder Checklist for DSM-5

OTHER OUTCOMES:
Acceptability | Immediate post-intervention
  The Insomnia Treatment Acceptability Scale-Behavioral Subscale
Participant Satisfaction | Change from immediately post-intervention satisfaction to one-month
  Client Satisfaction Questionnaire-8
Sleep Knowledge | During the intervention, immediately after baseline
  Sleep Scholar Quizzes
Average Nap Duration | Change from average one week Nap Duration at two weeks, three weeks, and four weeks
  The Consensus Sleep Diary; seven daily sleep diaries
Average Variance in Wake-Up Time | Change from average one week Variance in Wake-Up Time at two weeks, three weeks, and four weeks
  The Consensus Sleep Diary; seven daily sleep diaries
Average Variance in Time in Bed | Change from average one week Variance in Time in Bed at two weeks, three weeks, and four weeks
  The Consensus Sleep Diary; seven daily sleep diaries
Average Time from Bedtime to Trying to Sleep and From Wake Time to Rise Time | Change from average one week Time from Bedtime to Trying to Sleep and From Wake Time to Rise Time at two weeks, three weeks, and four weeks
  The Consensus Sleep Diary; seven daily sleep diaries

CONTACTS AND LOCATIONS:
Locations (1):
- Auburn University, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zuromski KL, Cero I, Witte TK. Insomnia symptoms drive changes in suicide ideation: A latent difference score model of community adults over a brief interval. J Abnorm Psychol. 2017 Aug;126(6):739-749. doi: 10.1037/abn0000282. Epub 2017 May 29. PMID 28557509
- [Background] Liu RT, Steele SJ, Hamilton JL, Do QBP, Furbish K, Burke TA, Martinez AP, Gerlus N. Sleep and suicide: A systematic review and meta-analysis of longitudinal studies. Clin Psychol Rev. 2020 Nov;81:101895. doi: 10.1016/j.cpr.2020.101895. Epub 2020 Aug 8. PMID 32801085
- [Background] Batterham PJ, Christensen H, Mackinnon AJ, Gosling JA, Thorndike FP, Ritterband LM, Glozier N, Griffiths KM. Trajectories of change and long-term outcomes in a randomised controlled trial of internet-based insomnia treatment to prevent depression. BJPsych Open. 2017 Sep 25;3(5):228-235. doi: 10.1192/bjpo.bp.117.005231. eCollection 2017 Sep. PMID 28959453
- [Background] Christensen H, Batterham PJ, Gosling JA, Ritterband LM, Griffiths KM, Thorndike FP, Glozier N, O'Dea B, Hickie IB, Mackinnon AJ. Effectiveness of an online insomnia program (SHUTi) for prevention of depressive episodes (the GoodNight Study): a randomised controlled trial. Lancet Psychiatry. 2016 Apr;3(4):333-41. doi: 10.1016/S2215-0366(15)00536-2. Epub 2016 Jan 28. PMID 26827250
- [Background] Thorndike FP, Saylor DK, Bailey ET, Gonder-Frederick L, Morin CM, Ritterband LM. Development and Perceived Utility and Impact of an Internet Intervention for Insomnia. E J Appl Psychol. 2008;4(2):32-42. doi: 10.7790/ejap.v4i2.133. PMID 20953264
- [Background] Ellis JG, Cushing T, Germain A. Treating Acute Insomnia: A Randomized Controlled Trial of a "Single-Shot" of Cognitive Behavioral Therapy for Insomnia. Sleep. 2015 Jun 1;38(6):971-8. doi: 10.5665/sleep.4752. PMID 25515106
- [Background] Downs MF, Eisenberg D. Help seeking and treatment use among suicidal college students. J Am Coll Health. 2012;60(2):104-14. doi: 10.1080/07448481.2011.619611. PMID 22316407
- [Background] Stinson K, Tang NK, Harvey AG. Barriers to treatment seeking in primary insomnia in the United Kingdom: a cross-sectional perspective. Sleep. 2006 Dec;29(12):1643-6. doi: 10.1093/sleep/29.12.1643. PMID 17252896
- [Background] Taylor DJ, Bramoweth AD, Grieser EA, Tatum JI, Roane BM. Epidemiology of insomnia in college students: relationship with mental health, quality of life, and substance use difficulties. Behav Ther. 2013 Sep;44(3):339-48. doi: 10.1016/j.beth.2012.12.001. Epub 2012 Dec 19. PMID 23768662
- [Background] Substance Abuse and Mental Health Services Administration. (2020). Key substance use and mental health indicators in the United States: Results from the 2019 National Survey on Drug Use and Health (HHS Publication No. PEP20-07-01-001, NSDUH Series H-55). 114.
- [Background] Substance Abuse and Mental Health Services Administration, Hedden, S. L., Kennet, J., Lipari, R., Medley, G., Tice, P., Copello, E. A. P., & Kroutil, L. A. (2015). Key Substance Use and Mental Health Indicators in the United States: Results from the 2015 National Survey on Drug Use and Health. 74.
- [Background] Pigeon WR, Funderburk JS, Cross W, Bishop TM, Crean HF. Brief CBT for insomnia delivered in primary care to patients endorsing suicidal ideation: a proof-of-concept randomized clinical trial. Transl Behav Med. 2019 Nov 25;9(6):1169-1177. doi: 10.1093/tbm/ibz108. PMID 31271210
- [Background] Pigeon WR, Funderburk J, Bishop TM, Crean HF. Brief cognitive behavioral therapy for insomnia delivered to depressed veterans receiving primary care services: A pilot study. J Affect Disord. 2017 Aug 1;217:105-111. doi: 10.1016/j.jad.2017.04.003. Epub 2017 Apr 6. PMID 28395207
- [Background] Hurst CS, Baranik LE, Daniel F. College student stressors: a review of the qualitative research. Stress Health. 2013 Oct;29(4):275-85. doi: 10.1002/smi.2465. Epub 2012 Oct 1. PMID 23023893
- [Background] Sexton-Radek K, Hartley A. College residential sleep environment. Psychol Rep. 2013 Dec;113(3):903-7. doi: 10.2466/06.10.PR0.113x27z2. PMID 24693819
- [Background] Gradisar M, Wolfson AR, Harvey AG, Hale L, Rosenberg R, Czeisler CA. The sleep and technology use of Americans: findings from the National Sleep Foundation's 2011 Sleep in America poll. J Clin Sleep Med. 2013 Dec 15;9(12):1291-9. doi: 10.5664/jcsm.3272. PMID 24340291
- [Background] Adams, S. K., Williford, D. N., Vaccaro, A., Kisler, T. S., Francis, A., & Newman, B. (2017). The young and the restless: Socializing trumps sleep, fear of missing out, and technological distractions in first-year college students. International Journal of Adolescence and Youth, 22(3), 337-348. https://doi.org/10.1080/02673843.2016.1181557
- [Background] Forquer LM, Camden AE, Gabriau KM, Johnson CM. Sleep patterns of college students at a public university. J Am Coll Health. 2008 Mar-Apr;56(5):563-5. doi: 10.3200/JACH.56.5.563-565. PMID 18400669
- [Background] Roepke SE, Duffy JF. Differential impact of chronotype on weekday and weekend sleep timing and duration. Nat Sci Sleep. 2010 Sep 1;2010(2):213-220. doi: 10.2147/NSS.S12572. PMID 20890372
- [Background] Sivertsen B, Pallesen S, Friborg O, Nilsen KB, Bakke OK, Goll JB, Hopstock LA. Sleep patterns and insomnia in a large population-based study of middle-aged and older adults: The Tromso study 2015-2016. J Sleep Res. 2021 Feb;30(1):e13095. doi: 10.1111/jsr.13095. Epub 2020 May 29. PMID 32469116
- [Background] Sivertsen B, Vedaa O, Harvey AG, Glozier N, Pallesen S, Aaro LE, Lonning KJ, Hysing M. Sleep patterns and insomnia in young adults: A national survey of Norwegian university students. J Sleep Res. 2019 Apr;28(2):e12790. doi: 10.1111/jsr.12790. Epub 2018 Dec 4. PMID 30515935
- [Background] Trockel M, Karlin BE, Taylor CB, Brown GK, Manber R. Effects of cognitive behavioral therapy for insomnia on suicidal ideation in veterans. Sleep. 2015 Feb 1;38(2):259-65. doi: 10.5665/sleep.4410. PMID 25515115
- [Background] Pigeon WR, Pinquart M, Conner K. Meta-analysis of sleep disturbance and suicidal thoughts and behaviors. J Clin Psychiatry. 2012 Sep;73(9):e1160-7. doi: 10.4088/JCP.11r07586. PMID 23059158
- [Background] Pigeon WR, Campbell CE, Possemato K, Ouimette P. Longitudinal relationships of insomnia, nightmares, and PTSD severity in recent combat veterans. J Psychosom Res. 2013 Dec;75(6):546-50. doi: 10.1016/j.jpsychores.2013.09.004. Epub 2013 Oct 2. PMID 24290044
- [Background] Blanco C, Okuda M, Wright C, Hasin DS, Grant BF, Liu SM, Olfson M. Mental health of college students and their non-college-attending peers: results from the National Epidemiologic Study on Alcohol and Related Conditions. Arch Gen Psychiatry. 2008 Dec;65(12):1429-37. doi: 10.1001/archpsyc.65.12.1429. PMID 19047530
- [Background] Smyth JM, Hockemeyer JR, Heron KE, Wonderlich SA, Pennebaker JW. Prevalence, type, disclosure, and severity of adverse life events in college students. J Am Coll Health. 2008 Jul-Aug;57(1):69-76. doi: 10.3200/JACH.57.1.69-76. PMID 18682348
- [Background] Hertenstein E, Feige B, Gmeiner T, Kienzler C, Spiegelhalder K, Johann A, Jansson-Frojmark M, Palagini L, Rucker G, Riemann D, Baglioni C. Insomnia as a predictor of mental disorders: A systematic review and meta-analysis. Sleep Med Rev. 2019 Feb;43:96-105. doi: 10.1016/j.smrv.2018.10.006. Epub 2018 Nov 16. PMID 30537570
- [Background] Geiger-Brown JM, Rogers VE, Liu W, Ludeman EM, Downton KD, Diaz-Abad M. Cognitive behavioral therapy in persons with comorbid insomnia: A meta-analysis. Sleep Med Rev. 2015 Oct;23:54-67. doi: 10.1016/j.smrv.2014.11.007. Epub 2014 Nov 29. PMID 25645130
- [Background] Seyffert M, Lagisetty P, Landgraf J, Chopra V, Pfeiffer PN, Conte ML, Rogers MA. Internet-Delivered Cognitive Behavioral Therapy to Treat Insomnia: A Systematic Review and Meta-Analysis. PLoS One. 2016 Feb 11;11(2):e0149139. doi: 10.1371/journal.pone.0149139. eCollection 2016. PMID 26867139
- [Background] Ye YY, Chen NK, Chen J, Liu J, Lin L, Liu YZ, Lang Y, Li XJ, Yang XJ, Jiang XJ. Internet-based cognitive-behavioural therapy for insomnia (ICBT-i): a meta-analysis of randomised controlled trials. BMJ Open. 2016 Nov 30;6(11):e010707. doi: 10.1136/bmjopen-2015-010707. PMID 27903557
- [Background] Ye YY, Zhang YF, Chen J, Liu J, Li XJ, Liu YZ, Lang Y, Lin L, Yang XJ, Jiang XJ. Internet-Based Cognitive Behavioral Therapy for Insomnia (ICBT-i) Improves Comorbid Anxiety and Depression-A Meta-Analysis of Randomized Controlled Trials. PLoS One. 2015 Nov 18;10(11):e0142258. doi: 10.1371/journal.pone.0142258. eCollection 2015. PMID 26581107
- [Background] Edinger JD, Arnedt JT, Bertisch SM, Carney CE, Harrington JJ, Lichstein KL, Sateia MJ, Troxel WM, Zhou ES, Kazmi U, Heald JL, Martin JL. Behavioral and psychological treatments for chronic insomnia disorder in adults: an American Academy of Sleep Medicine clinical practice guideline. J Clin Sleep Med. 2021 Feb 1;17(2):255-262. doi: 10.5664/jcsm.8986. PMID 33164742
- [Background] Edinger JD, Wohlgemuth WK, Radtke RA, Coffman CJ, Carney CE. Dose-response effects of cognitive-behavioral insomnia therapy: a randomized clinical trial. Sleep. 2007 Feb;30(2):203-12. doi: 10.1093/sleep/30.2.203. PMID 17326546
- [Background] Bootzin, Richard R., & Perlis, M. L. (2011). Stimulus control therapy. In M. Perlis, M. S. Aloia, & B. Khun (Eds.), Behavioral Treatments for Sleep Disorders (pp. 21-30). Elsevier.
- [Background] Bootzin, Richard R. (1972). Stimulus control treatment for insomnia. Proceedings of the American Psychological Association, 7, 395-396.
- [Background] Spielman, A. J., Yang, C.-M., & Glovinsky, P. B. (2016). Insomnia: Sleep Restriction Therapy. In M. Sateia & D. Buysse (Eds.), Insomnia: Diagnosis and Treatment (pp. 277-289).
- [Background] Oinas-Kukkonen, H., & Harjumaa, M. (2009). Persuasive Systems Design: Key Issues, Process Model, and System Features. Communications of the Association for Information Systems, 24. https://doi.org/10.17705/1CAIS.02428